CLINICAL TRIAL: NCT00490347
Title: Evaluation of the VentrAssistTM Left Ventricular Assist Device as a Bridge to Cardiac Transplantation - Feasibility Trial
Brief Title: VentrAssistTM LVAD as a Bridge to Cardiac Transplantation - Feasibility Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ventracor (Industry)
Collaborators: International Center for Health Outcomes and Innovation Research (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP070012
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: End-Stage Heart Failure; Cardiomyopathies
Keywords: VentrAssistTM; LVAD; End-stage heart failure; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: VentrAssist Left Ventricular Assist Device

SUMMARY:
The purpose of this trial is to determine the safety and feasibility of the VentrAssist LVAD in providing circulatory support for patients who require an LVAD as a bridge to cardiac transplantation.

ELIGIBILITY:
Inclusion Criteria (The following are general criteria; more specific criteria are included in the study protocol):

* Approved and listed for cardiac transplantation.
* Patient for whom LVAD implantation is planned as a clinically indicated bridge to cardiac transplantation.

Exclusion Criteria(The following are general criteria; more specific criteria are included in the study protocol):

* Presence of heart conditions that would contraindicate LVAD implantation by adversely affecting patient survival or LVAD function.
* Primary coagulopathy or platelet disorder; contraindication to anticoagulant or anti-platelet agents.
* Presence of any mechanical circulatory support other than intra-aortic balloon pump.
* Therapy with an investigational intervention at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-07; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
Quality of life
Functional status
Neurocognitive function

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Maryland Medical Center - Baltimore, Baltimore, Maryland
  - University of Minnesota Medical Center - Fairview, Minneapolis, Minnesota
  - New York Presbyterian Medical Center - Columbia, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania